CLINICAL TRIAL: NCT07372378
Title: Association of Various Introperative Tidal Volumes and Postoperative Pulmonary Complications After Video-assisted Thoracic Surgery
Brief Title: Association of Different Tidal Volumes and Postoperative Pulmonary Complications
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, xiangming fang, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: VolumePPC
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Complications; Hypoxemia During Surgery; Thoracic Surgery, Video Assisted; One Lung Ventillation (OLV); Lung Cancer (Non-Small Cell)
Keywords: pulmonary complications; hypoxemia; video-assisted thoracic surgery; one lung ventilation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of lung cancer in China is increasing year by year. Currently, the treatment primarily based on video-assisted thoracoscopic surgery (VATS) is still considered the optimal approach for early-stage non-small cell lung cancer. The widespread application of traditional one-lung ventilation (OLV) technology not only achieves effective lung isolation, but also facilitates exposure of the surgical field during thoracoscopic surgery, making it more convenient for surgeons to operate. However, the occurrence of hypoxemia during one-lung ventilation may pose a risk to patient safety.

One-lung ventilation can lead to increased intrapulmonary shunt, ventilation/perfusion (V/Q) mismatch, and ischemic-hypoxic lung injury. Hypoxemia is the major problem during one-lung ventilation. Postoperative pulmonary complications (PPCs) are among the major complications following thoracic and general anesthesia surgeries, including atelectasis, pneumonia, and respiratory failure, which significantly prolong hospital stay and increase mortality.

Low tidal volume lung-protective ventilation strategies have been widely implemented. Additionally, permissive hypercapnia, reducing peak airway pressure to minimize barotrauma, and decreasing FiO₂ all help reduce pulmonary complications.Recently, researchers have focused on optimizing ventilation strategies during OLV, such as using PEEP or low VT ventilation alone or in combination, or exploring different combinations of tidal volume and respiratory frequency under consistent minute ventilation (VE), aiming to balance lung protection and oxygenation, reduce complications, and improve patient outcomes.

However, to date, there is still no gold standard tidal volume ventilation strategy for reducing pulmonary complications in patients undergoing lung resection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years.
* ASA physical status I-II.
* The cardiopulmonary and other vital organ functions are basically normal, and the patient is able to tolerate surgery.
* Ariscat score > 26.
* Informed consent has been obtained.

Exclusion Criteria:

* Patients who refuse to participate in the clinical trial, or have cognitive impairment or impaired ability to understand and express themselves.
* ASA physical status ≥ III.
* Patients with congestive heart failure, severe aortic stenosis, or extensive pleural adhesions.
* Patients with severe psychiatric disorders or allergy to anesthesia-related medications.
* Patients with severe organ dysfunction such as the liver or kidney dysfunction.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing video-assisted lung surgery
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pulmonary Complications (PPCs) | 1-7 days after surgery
  Postoperative Pulmonary Complications (PPCs): Incidence of any PPC within 7 days postoperatively

SECONDARY OUTCOMES:
Incidence of hypoxemia | during surgery
  Incidence of hypoxemia: Occurring before the end of surgery
Length of Hospital Stay | through study completion, an average of 1 year
  Length of Hospital Stay

OTHER OUTCOMES:
Intraoperative Oxygenation Index | during surgery
  Intraoperative Oxygenation Index
Intraoperative Lung Compliance | during surgery
  Intraoperative Lung Compliance
Intraoperative Driving Pressure | during surgery
  Intraoperative Driving Pressure
Intraoperative Dead Space to Tidal Volume Ratio (Vd/Vt) | during surgery
  Intraoperative Dead Space to Tidal Volume Ratio (Vd/Vt)
Surgeon Satisfaction | At the end of surgery
  The degree of surgeon satisfaction regarding the performance, effectiveness, and experience of a procedure. A 10-point scale is used, 0 indicates complete dissatisfaction and 10 indicates complete satisfaction.
In-hospital mortality | through study completion, an average of 1 year
  In-hospital mortality
28-day mortality | 28 day postoperatively
  28-day mortality
90-day mortality | 90 day postoperatively
  90-day mortality

IPD SHARING:
Plan to Share IPD: No